CLINICAL TRIAL: NCT04573257
Title: Relationship Between Arteriosclerosis and Myocardial Work in Hypertensive Patients With Left Ventricular Ejection Fraction Retention
Brief Title: Effect of Aterial Stiffness on Myocardial Work in Patients With Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dongying Zhang, professor, Chongqing Medical University
Other Study IDs: 20200910
Record Dates: First submitted 2020-09-21; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Hypertension; Heart Disease, Hypertensive
Keywords: two-dimensional speckle tracking; hypertension; aterosclerosis; myocardial work
MeSH Terms: conditions — Hypertension; Heart Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- normotensive group: The medical history and basic examination and examination information were collected. Echocardiography including conventional cardiac ultrasound, tissue Doppler and two-dimensional speckle tracking to measure myocardial strain and noninvasive myocardial work were carried out , and the brachial-ankle pulse wave velocity was measured in parallel.
  Interventions: Other: Echocardiography and pulse wave velocity measurement
- Prehypertension group: The medical history and basic examination and examination information were collected. Echocardiography including conventional cardiac ultrasound, tissue Doppler and two-dimensional speckle tracking to measure myocardial strain and noninvasive myocardial work were carried out , and the brachial-ankle pulse wave velocity was measured in parallel.
  Interventions: Other: Echocardiography and pulse wave velocity measurement
- hypertensive group: The medical history and basic examination and examination information were collected. Echocardiography including conventional cardiac ultrasound, tissue Doppler and two-dimensional speckle tracking to measure myocardial strain and noninvasive myocardial work were carried out , and the brachial-ankle pulse wave velocity was measured in parallel.
  Interventions: Other: Echocardiography and pulse wave velocity measurement

INTERVENTIONS:
Other: Echocardiography and pulse wave velocity measurement — Echocardiography(Conventional ultrasonic imaging,tissue Doppler imaging and non invasive myocardial work) and pulse wave velocity measurement

SUMMARY:
Hypertension is a serious threat to human health and a major global economic burden.Chronic hypertension can cause left ventricular remodeling and loss of function, eventually leading to heart failure.Exploring the early changes and mechanisms of left ventricular cardiac function caused by hypertension, and to identify individuals who may develop into serious heart injury, may play a positive role in the early prevention and control of heart failure caused by hypertension.Therefore, this study intend to use two-dimensional speckle tracking technology, a non-invasive method to measure left ventricular pressure-strain loop to quantitatively reflect cardiac work index , to study different hypertension patients with normal left ventricular ejection fraction the change of the global and local cardiac work, and the influence of aterosclerosis in thes patients to myocardial work, and explore their relationship with ventricular remodeling and abnormal diastolic function.To improve the understanding of the pathophysiology of hypertension, hypertensive heart disease and heart failure, and to provide scientific support for the early prevention and control of such diseases.

DETAILED DESCRIPTION:
Hypertension is a serious threat to human health and a major global economic burden.Chronic hypertension can cause left ventricular remodeling and loss of function, eventually leading to heart failure. Ventricular remodeling in hypertensive patients is an adaptive and decompensating response to persistent elevated blood pressure and increased myocardial work load. Exploring the early changes and mechanisms of left ventricular cardiac function caused by hypertension, and to identify individuals who may develop into serious heart injury, may play a positive role in the early prevention and control of heart failure caused by hypertension.Therefore, this study intend to use two-dimensional speckle tracking technology, a non-invasive method to measure left ventricular pressure-strain loop to quantitatively reflect cardiac work index , to study different hypertension patients with normal left ventricular ejection fraction (including hypertension without heart damage performance with different degree of high blood pressure, hypertension with diastolic dysfunction , hypertension with left ventricular hypertrophy ) the change of the global and local cardiac work, and the influence of aterosclerosis in thes patients to myocardial work, and explore their relationship with ventricular remodeling and abnormal diastolic function.To improve the understanding of the pathophysiology of hypertension, hypertensive heart disease and heart failure, and to provide scientific support for the early prevention and control of such diseases.

ELIGIBILITY:
Inclusion Criteria:

Age 18-65 years

The diagnostic criteria of hypertension were blood pressure systolic blood pressure ≥140mmHg and/or diastolic blood pressure ≥90mmHg in the clinic or receiving antihypertensive drug treatment

The normal high-value diagnostic criteria for hypertension were systolic blood pressure 130-139mmhg and or diastolic blood pressure 85-90mmhg in the clinic

LVEF > 50%

Exclusion Criteria:

coronary atherosclerotic heart disease or symptoms of angina

Cardiomyopathy

Valvular heart disease

Diabetes

Atrial fibrillation

Renal function damage

Pregnancy

Secondary hypertension

Chemotherapy for malignant tumors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hypertension patients evaluated by echocardiography in theEchocardiography Center of the First Affiliated Hospital of Chongqing Medical University from September 2020 to January 2021.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
myocardial work | 2020.09-2021.01
  myocardial work measured by non-invasive left ventricular pressure-strain loop（2D speckle tracking echocardiography method by using the GE Vivid E95 ultrasound system ）

SECONDARY OUTCOMES:
brachial-ankle pulse wave velocity | 2020.09-2021.01
  brachial-ankle pulse wave velocity measured by OMRON BP-203RPEIII arteriosclerosis detector

CONTACTS AND LOCATIONS:
Overall Officials: QIN DUAN, Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, China

REFERENCES:
- [Derived] Duan Q, Ge P, Tao Y, Liao KL, Yang Y, Dong Q. Correlation between Ventricular-Arterial Coupling and Global Longitudinal Strain in Hypertensive With Preserved Ejection Fraction. Am J Hypertens. 2025 Oct 14:hpaf153. doi: 10.1093/ajh/hpaf153. Online ahead of print. PMID 41092222